CLINICAL TRIAL: NCT01016080
Title: Glutathione as an Oral Whitening Agent: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Role of Oral Glutathione in Skin Whitening
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Pravit Asawanonda, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COA840/2008
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Skin Whitening
Keywords: glutathione; melanin; whitening; UV spots; skin pigment
MeSH Terms: conditions — Pigmentation Disorders | interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral glutathione (Active Comparator): glutathione, 500 mg, taken orally twice daily
  Interventions: Drug: glutathione
- placebo capsules (Placebo Comparator): identical-appearing placebo capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: glutathione — 250 mg capsules, twice daily, orally
  Arms: oral glutathione
Drug: placebo — 250 mg capsules, twice daily, orally
  Arms: placebo capsules

SUMMARY:
Oral and intravenous glutathione have been used widely to whiten the skin. The investigators tested this hypothesis by giving oral glutathione for 4 weeks to medical students.

ELIGIBILITY:
Inclusion Criteria:

* Healthy medical students

Exclusion Criteria:

* history of skin cancer, especially melanoma
* consumption of any preparations containing glutathione within 1 month of enrollment
* pigmentary disorders or any dermatoses

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Skin melanin index | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand